CLINICAL TRIAL: NCT05116293
Title: Effect of Gender-Affirming Testosterone Therapy on Drug Metabolism, Transport, and Gut Microbiota
Brief Title: Effect of Testosterone Treatment on Drug Metabolism and Transport
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lauren Cirrincione, Assistant Professor, Pharmacy, University of Washington
Other Study IDs: STUDY00011644
Record Dates: First submitted 2021-10-15; First posted 2021-11-11 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Transgender Persons
Keywords: Testosterone Treatment
MeSH Terms: interventions — Midazolam; Digoxin; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Midazolam oral solution — Oral syrup
Drug: Digoxin Oral Tablet — Oral tablet
Drug: Acetaminophen Oral Tablet — Oral tablet

SUMMARY:
This project will evaluate the effect of gender-affirming testosterone treatment on how other medications are processed by the body.

DETAILED DESCRIPTION:
Gender-affirming hormone therapy may include testosterone, a hormone that the body creates and uses naturally. Testosterone is prepared as a medication that patients may take to increase hormone levels. Changes in testosterone concentrations in the body may affect how the body processes other medicines. The purpose of this study is to find out how testosterone therapy affects a single tracer dose of approved medicines in the blood (midazolam, digoxin, and acetaminophen) and to confirm testosterone treatment does not affect natural bacterial in the gut.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified trans* adult at least 18 years of age.
* Not taking testosterone treatment currently.
* Planning to start testosterone treatment through care provider for gender-affirming medical care.

Exclusion Criteria:

* Unwilling/unable to return for project follow-up visits.
* Unwilling/unable to provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as transgender or trans nonbinary
Study Population: Transgender adults planning to take testosterone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
midazolam AUC ratio (treatment/control) | 0-48 hours
  ratio of the area under of the plasma concentration time curve (AUC) of midazolam in the presence to absence of gender-affirming testosterone treatment.

SECONDARY OUTCOMES:
midazolam Cmax ratio (treatment/control) | 0-48 hours
  ratio of the maximum plasma concentration (Cmax) of midazolam in the presence to absence of gender-affirming testosterone treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Cirrincione, MPH,Pharm D, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States